CLINICAL TRIAL: NCT00472069
Title: EVALUATION Of A NEW THERAPEUTIC STRATEGY FOR URETHRAL SPHINCTER INSUFFICIENCY BASED ON THE INTRA-URETHRAL IMPLANTATION OF AUTOLOGOUS MYOFIBERS WITH THEIR SATELLITE CELLS
Brief Title: A New Therapeutic Strategy for Urethral Sphincter Insufficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Cecile KEDZIA, Department Clinical Research of developpement
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P060505
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2007-09

CONDITIONS: Stress Urinary Incontinence; Urethral Intrinsic Sphincter Deficiency
Keywords: Stress Urinary Incontinence; striated urethral sphincter insufficiency; myofibers; satellite cells; myotubes; urethral; Muscle fibres
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): transplantation of the squeletic muscular cells
  Interventions: Procedure: transplantation of the squeletic muscular cells

INTERVENTIONS:
Procedure: transplantation of the squeletic muscular cells — transplantation of the squeletic muscular cells

SUMMARY:
Stress urinary incontinence is a frequent condition that can be caused by urethral sphincter insufficiency and results in a dramatic deterioration of the quality of life. We developed a new therapeutic strategy for stress urinary incontinence based on the implantation myofibers with their satellite cells in the urethra. The aim of this procedure is to generate functional tissue acting like a new sphincter in the urethra

DETAILED DESCRIPTION:
stress urinary incontinence is a frequent condition that can be caused by urethral sphincter insufficiency and results in a dramatic deterioration of the quality of life. We developed a new therapeutic strategy for stress urinary incontinence based on the implantation myofibers with their satellite cells. The principle of this procedure relies on the activation in vivo of the satellite cells present around each myofibers. Satellite cell activation is concomitant with myofiber death that occurs after their implantation. Activated satellite proliferate and fuse to form myotubes replacing the parental myofibers thus leading to the reconstitution of the muscle mass that was initially implanted. Preliminary studies in the pig showed the regenerated muscle tissue in the urethra was innervated by urethral nerves and developed tonic contractions acting like a new sphincter. This procedure does not include a phase of satellite cell amplification ex vivo, as standard methods of satellite cell transfer, and rather relies on the natural myogenic capacities of these cells. Thus, the procedure of cell transfer into the urethra is considerably simplified and can be performed in one step in the operating room.This therapeutic strategy could represent an alternative to the artificial urinary sphincter.

ELIGIBILITY:
Inclusion Criteria:

* Men or women from 40 to 75 years old, suffering from urinary incontinence since at least 6 months and candidate for a surgical treatment (artificial urinary sphincter, synthetic compressive tapes or adjustable balloons).

The myofiber implantation procedure will be proposed after failure of pelvic floor exercises.

* The observation of urine leakage during cough in consultation or during urodynamic (with absence of abnormal vesical contraction) and a score MHU > 2 (domain of stress urinary incontinence) will be considered as the main diagnostic criteria.
* An urethral closure pressure lower than 40 cm H20 will be the main urodynamic diagnostic criterion
* For women: a negative BONNEY test, and Qtip test<40° (c.f. annex) demonstrating the absence of vesica-urethral hypermobility.

  24 hours Pad test > 20g.

Exclusion Criteria:

* Incapacity to answer the questionnaires of evaluation.
* History of pelvic radiotherapy.
* Disorder of hemostasis.
* Untreated urinary infection.
* Genetically determined or acquired muscular disease.
* Neurological disorder (Parkinson's disease, multiple sclerosis, spina BIFIDA, medullary traumatism).
* The patients suffering from stress urinary incontinence due to vesica-urethral hypermobility (positive BONNEY test and Qtip test >40°) will not be included in the study because the referenced treatment is the implantation of a vaginal tape supporting the urethra.
* Incomplete vesical emptying. Residual volume > 20% of the urinated volume with a micturition >150cc.
* Dysuria: maximum urinary flow < 12 ml/sec, IPSS score>7 or score (men) or MHU dysuria domain none equal to 0 at woman.
* Vesical instability (bladder contraction > 10 cm H20 during the vesical filling of the cysto-manometry). bladder capacity (B3) < 300 DC.
* Urethral Stenosis (ureterocystoscopy).
* Previous surgeries for urinary incontinence do not constitute a criterion of exclusion.
* Pregnancy or intention of pregnancy throughout study. A test of pregnancy will be carried out with the visit of inclusion.
* Urethral diverticulum.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Clinical tolerance and feasibility of a new therapeutic strategy for stress urinary incontinence based on intra urethral myofiber implantation of autologous myofibers with their satellite cells | 3 months

SECONDARY OUTCOMES:
Effects of this treatment on urinary continence in order to consider a phase II later on. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: René YIOU, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Henri Mondor service Urologie, Créteil, France